CLINICAL TRIAL: NCT03285373
Title: Non-Interventional, Cross-sectional Study to Describe NOACs Management ss in Patients With Non-valvular Atrial Fibrillation (NVAF) in Spain.
Brief Title: This Study Observes the Use of New Oral Anticoagulants (NOACs) in Patients With a Heart Rhythm Disorder in Spain
Acronym: RE-CONOCE
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0287
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with NVAF: patients with Non Valvular Atrial Fibrillation
  Interventions: Drug: NOAC

INTERVENTIONS:
Drug: NOAC — New Oral Anticoagulant

SUMMARY:
The primary objective of the study is to describe the usage of NOACs in patients with NVAF, in the hospital setting, based on the baseline characteristics at the time of first NOAC initiation.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and provides written informed consent to participate in this study
* The patient is at least 18 years of age
* The patient has a diagnosis of non-valvular atrial fibrillation (NVAF)
* The patient is on treatment with NOAC according to its approved local SmPC and has initiated his first NOAC starting from November 2016

Exclusion Criteria:

-if the current participating patient participate in any clinical trial of a drug or device will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1.000 patients with NVAF currently on NOAC treatment and having initiated their first NOAC starting from November 2016 (Health Authorities positioning report publication) are planned to be included in the study. To minimize selection bias at the patient level, 10 consecutive patients from each site who meet entry criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1008 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Canals, +34607550925, Study Chair — mireia.canals@boehringer-ingelheim.com
Locations (74):
- Spain (74):
  - Clínica Modelo, A Coruña
  - Hospital Universatio de Albacete, Albacete
  - Hospital Quirónsalud Sur, Alcorcón (Madrid)
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Dr. José Molina Orosa, Arrecife, Las Palmas
  - H de Cabueñes, Asturias
  - Hospital Infanta Cristina, Badajoz
  - Clínica Sagrada Familia, Barcelona
  - Medical Practice, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - H. del Mar, Barcelona
  - Hospital del Mar, Barcelona
  - H. Residencia Sant Camil, Barcelona
  - H. Moisés Broggi, Barcelona
  - Hospital Basurto, Bilbao
  - H Aranda Duero, Burgos
  - Medical Practice, Castellon
  - Hospital de Cáceres, Cáceres
  - Medical Practice, Córdoba
  - Centro Médico Puerto, El Puerto de Santa Maria (Cádiz)
  - Hospital General de Elche, Elche (Alicante)
  - Hospital Vinalopo Salud, Elche (Alicante)
  - Hospital García Orcoyen, Estella (Navarra)
  - Clínica Del Río Estepona y San Pedro, Estepona (Málaga)
  - Complejo Hospitalario Arquitecto Marcide, Ferrol (A Coruña)
  - Hospital Galdakao, Galdakao (Vizcaya)
  - Medical Practice, Gandía (Valencia)
  - Hospital Vithas La Salud, Granada
  - Medical Practice, Granada
  - Medical Practice, Granollers (Barcelona)
  - H. U. Guadalajara, Guadalajara
  - Hospital Universitario de Bellvitge, Hospitalet de Ll (Barcelona)
  - Hospital Juan Ramon Jiménez, Huelva
  - Medical Practice, Huesca
  - H. Universitario Dr. Negrín, Las Palmas
  - Hospital General San Agustin, Linares (Jaen)
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital de la Princesa, Madrid
  - Hospital Nuestra Señora del Rosario, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - H. Quirón Salud H. Sur Alcorcón, Madrid
  - Hospital Universitario Puerta del Hierro, Majadahonda (Madrid)
  - Hospital de Manises, Manises (Valencia)
  - Hospital Ochoa, Marbella (Málaga)
  - Hospital de Mataró, Mataró (Barcelona)
  - Hospital de Mérida, Mérida
  - Hospital Universitario Central de Asturias, Oviedo (Asturias)
  - Hospital de Son Llatzer, Palma de Mallorca (Baleares)
  - Hospital Quirón Campo de Gibraltar, Palmones (Cádiz)
  - Centro de Especialidades Dr. San Martin, Pamplona
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitari Parc Taulí, Sabadell (Barcelona)
  - H. C. U. Salamanca, Salamanca
  - Policlínic Sant Cugat, Sant Cugat Del Valles (Barcelona)
  - Hospital Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Complejo H. Universitario de Canarias, Santa Cruz de Tenerife
  - CH Santiago de Compostela, Santiago de Compostela (A Coruña)
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela (A Coruña)
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela (A Coruña)
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Duque del Infantado, Seville
  - Medical Practice, Seville
  - Hospital Santa Santa Bárbara, Soria
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - HM Hospitales Madrid, Torrelodones (Madrid)
  - Clínica Santa Elena, Torremolinos
  - Pius Hospital de Valls, Valls (Tarragona)
  - Hospital Universitari de La Plana, Vila-Real (Castellón)
  - Hospital Lluis Alcanyis, Xàtiva (Valencia)
  - Complejo Asistencial de Zamora, Zamora
  - H. Clínico Universitario, Zaragoza
  - H. Miguel Servet, Zaragoza
  - H. Royo Villanova, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Non Valvular Atrial Fibrillation (NVAF) in Spain, mainly from the hospital setting were on treatment with New Oral Anticoagulant (NOAC) according to its approved local Summary of Product Characteristics (SmPC) and have initiated their first NOAC starting from November 2016 were included in this trial.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Subjects attended specialist sites in Spain to ensure that subjects met all incl/excl criteria. 45 patients (out of 1008 enrolled), did not meet at least one of the selection criteria and were considered not eligible. Data analysis was carried out with 963 eligible patients.
Groups:
- Dabigatran: Patients with Non Valvular Atrial Fibrillation (NVAF) started treatment with Dabigatran according to the SmPC.
- Rivaroxaban: Patients with Non Valvular Atrial Fibrillation (NVAF) started treatment with Rivaroxaban according to the SmPC.
- Apixaban: Patients with Non Valvular Atrial Fibrillation (NVAF) started treatment with Apixaban according to the SmPC.
- Edoxaban: Patients with Non Valvular Atrial Fibrillation (NVAF) started treatment with Edoxaban according to the SmPC.
Period: Overall Study
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban
Started | 314 | 253 | 266 | 130
Completed | 314 | 253 | 266 | 130
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria).
Groups:
- All Patients: Patients with Non Valvular Atrial Fibrillation (NVAF) started treatment with Dabigatran, Rivaroxaban, Apixaban or Edoxaban according to the SmPC from November2016 to January2019.
Arm/Group | All Patients
Number analyzed (Participants) | 963
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at baseline visit.
  Years | 73.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 406
  Male | 557
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Usage of NOAC Based on Baseline Characteristics: Age at the Time of the First NOAC Initiation
Description: Usage of NOAC in patients diagnosed with NVAF, in the hospital setting, based on the baseline characteristics; age, at the time of the start of the first NOAC initiation.
Time Frame: Start of the first NOAC treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | All Patients
Number analyzed (Participants) | 314 | 253 | 266 | 130 | 963
Years | 72.8 (9.9) | 72.5 (10.7) | 72.6 (9.8) | 74.0 (10.0) | 72.8 (10.1)

2. Primary Outcome: Usage of NOAC Based on Baseline Characteristics: CHA2DS2-VASc Scores at the Time of the First NOAC Initiation
Description: Usage of NOAC in patients diagnosed with NVAF, in the hospital setting, based on the baseline characteristics: Congestive heart failure, Hypertension, Age (> 75), Diabetes mellitus, Stroke/TIA, Vascular disease, Age 65-74, Sex Category (CHA2DS2-VASc Score) at the time of the start of the first NOAC initiation.
  The CHA2DS2-VASc score is a clinical prediction rule to estimate the risk of stroke in patients with Atrial Fibrillation (AF); it is frequently used to determine the need for an anticoagulation therapy, relating the high scores to a great risk of stroke and a low score corresponds to a lower risk of stroke. CHA2DS2-VASc stroke risk score may range from 0 to 9 with 0 being the best outcome.
Time Frame: Start of the first NOAC treatment
Population: The analysis population consisted of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria). For 21 patients CHA2DS2-VASc score was not available.
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | All Patients
Number analyzed (Participants) | 308 | 251 | 254 | 129 | 942
Unit on Scale | 3.2 (1.5) | 3.3 (1.6) | 3.3 (1.5) | 3.3 (1.5) | 3.3 (1.5)

3. Primary Outcome: Number of Patients on Risk Based on CHA2DS2-VASc Scores at the Time of the First NOAC Initiation
Description: Number of patients on risk (Low, Moderate and High) based on CHA2DS2-VASc Scores at the time of the start of the first NOAC initiation.
  The total CHA2DS2-VASc Scores score was stratified by category according to the following classification:
  1. Low risk (score 0 in male; score 1 in female)
  2. Moderate risk (score 1 in male; score 2 in female)
  3. High risk (score ≥2 in male; score ≥3 in female)
Time Frame: Start of the first NOAC treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | All Patients
Number analyzed (Participants) | 308 | 251 | 254 | 129 | 942
Participants
  Low risk | 3 | 10 | 3 | 0 | 16
  Moderate risk | 53 | 34 | 36 | 21 | 144
  High risk | 252 | 207 | 215 | 108 | 782

4. Primary Outcome: Usage of NOAC Based on Baseline Characteristics: HAS-BLED Score at the Time of the First NOAC Initiation
Description: Usage of NOAC in patients diagnosed with NVAF, in the hospital setting, based on the baseline characteristics: Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile INR, Elderly (>65 years), Drugs and Alcohol (HAS-BLED Score) at the time of the start of the first NOAC initiation. HAS-BLED bleeding risk score may range from 0 to 9 with 0 being the best outcome. The high scores to a great risk of bleeding and a low score corresponds to a lower risk of bleeding.
Time Frame: Start of the first NOAC treatment
Population: The analysis population consisted of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria). For 23 patients the HAS-BLED score was not available.
Measure: Mean (Standard Deviation); unit: unit on scale
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | All Patients
Number analyzed (Participants) | 308 | 251 | 253 | 128 | 940
unit on scale | 1.8 (1.0) | 1.8 (1.1) | 1.7 (1.1) | 1.8 (1.0) | 1.8 (1.1)

5. Primary Outcome: Number of Patients on Risk Based on HAS-BLED Score at the Time of the First NOAC Initiation
Description: Number of patients on risk (Low, Moderate and High) based on HAS-BLED Score at the time of the start of the first NOAC initiation.
  The total HAS-BLED Score was stratified by category according to the following classification:
  1. Low risk (score 0)
  2. Moderate risk (score 1-2)
  3. High risk (score ≥3)
Time Frame: Start of the first NOAC treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | All Patients
Number analyzed (Participants) | 308 | 251 | 253 | 128 | 940
Participants
  Low risk | 17 | 29 | 27 | 11 | 84
  Moderate risk | 219 | 157 | 170 | 86 | 632
  High risk | 72 | 65 | 56 | 31 | 224

6. Secondary Outcome: Appropriateness of NOACs Prescription
Description: Appropriateness of NOACs prescription based on national recommendations. For this, it was reviewed if the presence of at least one of the following clinical reason or reason related to International Normalized Ratio (INR) control were met.
  Reason 1: Patients with known hypersensitivity or with specific contraindications to the use of acenocoumarol or warfarin; Reason 2: Patients with a history of intracranial hemorrhage (ICH) (except during the acute phase); Reason 3: Patients with ischemic stroke who present high-risk clinical and neuroimaging criteria for ICH; Reason 4: Patients on VKA treatment who suffer from severe arterial thromboembolic events despite good INR control; Reason 5: Patients who have started treatment with VKA in which it is not possible to maintain INR control within range (2-3) despite good therapeutic compliance; Reason 6: impossibility of access to conventional INR control; Reason 7: Other reason; Reason 8; Unknown.
Time Frame: single visit (Day 1)
Population: The analysis population consisted of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria). As per protocol this endpoint was to be analysed for the entire eligible patients. Thus, this endpoint was not analysed by NOAC type.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 963
Participants
  Reason 1 | 88
  Reason 2 | 10
  Reason 3 | 16
  Reason 4 | 16
  Reason 5 | 271
  Reason 6 | 102
  Reason 7 | 342
  Reason 8 | 118

7. Secondary Outcome: Mean Number of Visits to the Physician Per Year
Description: Mean number of visits to the physician per year considered for the NOAC Management.
Time Frame: 1 year (data collected during single visit on day 1)
Population: The analysis population consisted of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria).As per protocol this endpoint was to be analysed for the entire eligible patients. Thus, this endpoint was not analysed by NOAC type.
Measure: Mean (Standard Deviation); unit: visits per year
Arm/Group | All Patients
Number analyzed (Participants) | 963
visits per year | 2.0 (1.1)

8. Secondary Outcome: Duration of First NOAC, All NOAC and Subsequent NOAC Treatment
Description: Duration of NOAC treatment (First NOAC, All NOAC and Subsequent NOAC).
Time Frame: Through the observational period with an average of 9.4 (first NOAC), 9.6 (All NOAC) and 5.1 (Subsequent NOAC) months, data collected during a single visit.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | All Patients
Number analyzed (Participants) | 963
Months
  First NOAC | 9.4 (6.5)
  All NOAC | 9.6 (6.5)
  Subsequent NOAC | 5.1 (4.1)

9. Secondary Outcome: Number of Patients Who Required Discontinuing the NOAC Treatment, to Adjust the NOAC Dose or to Change to a New NOAC
Description: Number of patients who required discontinuing the NOAC treatment, to adjust the NOAC dose or to change to a new NOAC
Time Frame: single visit (Day 1)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 963
Participants
  Discontinue treatment | 4
  Dose adjustment | 20
  Change to a new NOAC | 32
  No change | 907

10. Secondary Outcome: Number of Patients Who Changed From One NOAC to a New NOAC Type and Dose
Description: Number of patients who changed from one NOAC to a new NOAC type and dose. The treatment and its dose displayed below refer to the subsequent NOAC.
Time Frame: single visit (Day 1)
Population: The analysis population consisted of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria) who changed to a new NOAC. As per protocol this endpoint was to be analysed overall for all eligible patients who changed to a new NOAC. Thus, this endpoint was not analysed by NOAC type.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 32
Participants
  Dabigatran 110 mg | 5
  Dabigatran 150 mg | 4
  Rivaroxaban 10 mg | 1
  Rivaroxaban 15 mg | 2
  Rivaroxaban 20 mg | 4
  Apixaban 2.5 mg | 2
  Apixaban 5 mg | 8
  Edoxaban 30 mg | 2
  Edoxaban 60 mg | 4

11. Secondary Outcome: Reason for Treatment Changes
Description: Reason for treatment changes such as discontinuing the NOAC treatment, to adjust the NOAC dose or to change to a new NOAC.
Time Frame: Start of the first NOAC treatment
Population: The analysis population consisted of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria) who required treatment changes.As per protocol this endpoint was to be analysed overall for all eligible patients who required treatment changes. Thus, this endpoint was not analysed by NOAC type.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 56
Participants
  Lack of efficacy | 5
  Investigator decision | 30
  Patient decision | 7
  Adverse event | 14

12. Secondary Outcome: Number of Patients With Previous Treatment With Vitamin K Antagonists
Description: Number of patient with Previous Treatment with Vitamin K Antagonists.
Time Frame: single visit (Day 1)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | All Patients
Number analyzed (Participants) | 314 | 253 | 266 | 130 | 963
Participants
  Yes | 146 | 125 | 100 | 53 | 424
  No | 168 | 128 | 166 | 77 | 539

13. Secondary Outcome: Duration of Previous VKA Treatment
Description: Duration of previous VKA treatment is the time from start of the VKA treatment until stopped to start with the first NOAC
Time Frame: Through the observational period with an average of 43.8 months, data collected during a single visit.
Population: The analysis population consisted of all eligible patients (i.e. all patients fulfilling all inclusion criteria and no exclusion criteria). As per protocol this endpoint was to be analysed only for patients with previous VKA treatment (n=424). Dates of start and/or stop of previous VKA treatment were not available for 62 patients.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Edoxaban | All Patients
Number analyzed (Participants) | 124 | 107 | 81 | 50 | 362
Months | 46.6 (52.5) | 37.0 (50.6) | 54.5 (58.9) | 34.0 (47.9) | 43.8 (53.2)

14. Secondary Outcome: Patient's Knowledge About His Condition
Description: At the time of the inclusion, the physician performed a following small questionnaire to the patients, to answer yes/no, in order to assess the patient's knowledge about his illness and the anticoagulant treatment prescribed.
  Question 1. Do you know why you are being treated with an anticoagulant? Question 2. Do you know which the effect of the anticoagulant treatment is? Question 3. Do you know what could happen if you don't take the anticoagulant treatment? Question 4. Do you mind taking the anticoagulant treatment?
Time Frame: single visit (Day 1)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 963
Participants
  Question 1.: Yes | 845
  Question 1.: No | 118
  Question 2.: Yes | 820
  Question 2.: No | 143
  Question 3.: Yes | 766
  Question 3.: No | 197
  Question 4.: Yes | 333
  Question 4.: No | 630

ADVERSE EVENTS:
Time Frame: From Informed consent signed until the end of the trial, up to 12 months.
Description: The study design was of non-interventional nature and the study was conducted within the conditions of the approved marketing authorization. Sufficient data were available to support the evidence on the safety and efficacy of the studied BI drug. For this reason Adverse Drug Reactions (ADR) and fatal Adverse Events (AE) were only collected for one of the NOACs (dabigatran). No data was collected for the other NOACs (Rivaroxaban, Apixaban and Edoxaban) reported on in this study.
Arm/Group | Dabigatran
All-Cause Mortality (participants affected / at risk) | 1/314
Serious Adverse Events (participants affected / at risk) | 3/314
Other Adverse Events (participants affected / at risk) | 0/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran (N=314)
Sudden death (General disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT03285373/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03285373/SAP_001.pdf